CLINICAL TRIAL: NCT00777426
Title: HIV-1 Specific Immune Responses in Thai Individuals With HIV Dementia
Status: Completed | Type: Observational
Sponsor: SEARCH Research Foundation (Other)
Responsible Party: Principal Investigator, Assoc.Prof.Jintanat Ananworanich, M.D., Assoc.Prof.Jintanat Ananworanich, M.D., SEARCH Research Foundation
Other Study IDs: SEARCH 007
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: HIV Infections
Keywords: HIV positive with HAD
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PBMC, Plasma, Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Thai HAD individuals (25 cases)
- Thai Non-HAD individuals (25 cases)
- Thai Non-infected individuals (10 cases)

SUMMARY:
A total of 60 participants will be enrolled. They will be in 3 groups

1. ARV-naïve, HIV-positive ≥ 20 year of age with HAD (n=25) who intend to start ARV
2. ARV-naïve, HIV-positive ≥ 20 year of age without HAD (n=25), who intend to start ARV
3. HIV-negative ≥ 20 year of age (n=10). The protocol team will work with the primary care physician to ensure that the subjects receive standard HIV and ARV care; however, initiation of ARV is not a requirement of the study and ARV will not be provided by the study.

Participant accrual will include 10-15 participants per year. HIV-positive subjects will be tentatively enrolled in HAD vs. non-HAD groups by the enrolling neurologist and subsequently confirmed to that group by a consensus conference held every 6 months by the study neurologists. In cases of disagreement, cases will be re-assigned to the consensus conference determination and recruitment will continue. An external validation consensus conference will be conducted as well every 6-12 months to monitor correct assignment of the level of impairment.

DETAILED DESCRIPTION:
This application focuses on the role of cellular immune responses in HIV dementia (HAD) versus non-HAD individuals in a cognitively characterized cohort followed for one year.

Increasing evidence links strong CD4+ T helper function to robust CD8+ CTL responses. HIV-1-infected individuals who are able to maintain strong HIV-1 specific T cell responses have better clinical outcomes and rarely develop neurological signs or symptoms. Monocyte/macrophage (M/M) infiltration into the white matter of the brain is a hallmark of HAD; however, the mechanisms by which M/M are recruited to the brain are not clearly understood. We hypothesize that the loss of specific HIV-1 T cell response results in activation/dysregulation of M/M leading to their accumulation in the brain.

To test this hypothesis will characterize Thai HIV-1-infected individuals as follows: 25 HAD individuals, 25 CD4-, education-, gender-, and age-matched non-HAD individuals and 10 HIV negative controls. We will then: 1) define CD4+ and CD8+ T cell function by evaluating HIV-1 specific responses in HAD vs. non-HAD groups; 2) simultaneously correlate these responses to M/M subpopulation cell number, percentage, and immune function; 3) correlate these responses to HIV-1 proviral load and autologous viral sequences (viral escape sequences and HIV quasispecies); and 4) evaluate the impact of ARV on dementia related to changes in immunological responses. Since little is known of the interaction between CD4+ T helper responses, CTL function, and the level of M/M subpopulation activation in the neuropathogenesis of HAD, this innovative study will elucidate the role of HIV-1 specific immune responses in HAD and provide new insights into HIV-1 neuropathogenesis and its relationship to peripheral immune responses, potentially opening exciting new areas for further investigation.

ELIGIBILITY:
Inclusion Criteria:

Group Thai HAD individuals

* 20 years of age

  * not currently receiving nor have ever received antiretroviral medications
  * not explained by opportunistic infections or causes other than HIV on the basis of clinical assessment and neuropsychological testing and eligible for inclusion.

Group Thai Non-HAD individuals

* will be matched with a seropositive Thai patient with similar age (same decade), education (less than high school degree, high school degree +/- some college, college degree +), gender, and CD4 group
* HIV positive
* not currently receiving nor have ever received antiretroviral medications.

Group Thai Non-HAD individuals will be matched with a Thai seronegative patient by age (same decade), and education (less than high school degree, high school degree +/- some college, college degree+), and gender.

Exclusion Criteria:

* Head injury with loss of consciousness greater than 1 hour
* Current or past illicit drug use (less then 5 years) or positive drug screen for amphetamine, methamphetamines, cocaine, marijuana, or narcotics at either screening or entry.
* Inability to provide informed consent or lack of designated surrogate who can provide consent
* The following laboratory values:
* PT/PTT > the upper limit of normal (ULN) or INR > 1.1
* Hemoglobin < 9.0 mg/dL
* ALT > 5x ULN
* serum creatinine > 2x ULN or creatinine clearance < 30 cc per min by Cockroft-Gault formula
* Acute illness within 30 days prior to entry, persistent and active AIDS- defining opportunistic infection or autoimmune disease. Stable treated opportunistic infections on maintenance therapy, minor infections such as oral thrush and Kaposi's Sarcoma limited to the skin will be allowed.
* Current or recent fevers or meningeal signs suggestive of CNS opportunistic infection.*
* History of pre-existing neurologic disease to include stroke, multiple sclerosis
* History of psychiatric illness including schizophrenia, bipolar disorder, anxiety disorder, panic attacks, or post traumatic stress disorder. Patients with active major depression will be excluded as well - patients with past depression that is controlled and patients with or minor depressive symptoms will be allowed to enroll.
* Known learning disability including dyslexia.
* Positive Hepatitis C serology (Hepatitic C Ab)
* Confusion or other signs and symptoms of metabolic encephalopathy or delirium
* Mass consistent with opportunistic infection or tumor on CT or MRI of the head, or focal neurological deficit on examination consistent with possible brain lesion.*
* Other conditions that could explain neurocognitive decline in the opinion of the investigator such as hypothyroidism, vitamin B12 deficiency or neurosyphilis.
* Pregnancy.
* Not willing to take an MRI.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 60 participants will be enrolled. They will be in 3 groups
  1. ARV-naïve, HIV-positive ≥ 20 year of age with HAD (n=25) who intend to start ARV
  2. ARV-naïve, HIV-positive ≥ 20 year of age without HAD (n=25), who intend to start ARV
  3. HIV-negative ≥ 20 year of age (n=10). The protocol team will work with the primary care physician to ensure that the subjects receive standard HIV and ARV care; however, initiation of ARV is not a requirement of the study and ARV will not be provided by the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-09; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Assess the HIV-1 specific CD4+ T helper cell and CD8+ CTL responses in individuals with and without HAD prior to initiation of ARV | May 2013

SECONDARY OUTCOMES:
Measure M/M dysregulation/activation and correlate this with HIV-1 specific CD4+ and CD8+ T cell responses prior to initiation of ARV | May 2013
Correlate the impact of ARV on HAD with qualitative and quantitative changes in CD4+ and CD8+ HIV-1 specific responses | May 2013

CONTACTS AND LOCATIONS:
Overall Officials: Jintanat Ananworanich, MD, Study Chair — SEARCH Research Foundation
Locations (1):
- SEARCH Thailand, Bangkok, Bangkok, Thailand

REFERENCES:
- See also: South East Asia Research Collaboration with Hawaii (SEARCH) — http://www.searchthailand.org